CLINICAL TRIAL: NCT06820424
Title: A Phase I Clinical Study to Evaluate the Safety and Preliminary Efficacy of CDH17 CAR-T in Patients with CDH17-positive Advanced Solid Tumors
Brief Title: Safety and Preliminary Efficacy of Anti-CDH17 CAR-T Cell Therapy in Patients with CDH17-positive Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Collaborators: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-22-013
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: CDH17-positive Advanced Solid Tumors
Keywords: CDH17 CAR-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-CDH17 CAR-T cells (Experimental): CDH17 CAR-T is a novel CAR cell therapy for the treatment of advanced solid tumors.
  Interventions: Biological: Anti-CDH17 CAR-T cells infusion

INTERVENTIONS:
Biological: Anti-CDH17 CAR-T cells infusion — Subiects who meet the enrollment conditions will receive intravenous infusion of anti-CDH17 CAR-T Cells after lymphodepleting therapy.

SUMMARY:
This is a single-center, open-label, single-arm study to evaluate the safety and preliminary efficacy of anti-CDH17 CAR-T cells in patients with CDH17-positive advanced solid tumors.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm study to evaluate the safety and preliminary efficacy of anti-CDH17 CAR-T cells in patients with CDH17-positive advanced solid tumors.A leukapheresis procedure will be performed to manufacture Anti-CDH17 chimeric antigen receptor (CAR) modified T cells. Prior to Anti-CDH17 CAR-T cells infusion subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide. After infusion, the safety and efficacy of CAR-T therapy was evaluated by investigators.

ELIGIBILITY:
Inclusion Criteria:

1. The patient understands and voluntarily signs the informed consent form, and is expected to complete the follow-up examination and treatment of the study procedures;
2. Age 18-75 years old, gender unlimited;
3. Tumor patients who have positive expression of CDH17 target in tumor tissues measured by immunohistochemistry (IHC) in a laboratory approved by the partner, and have no standard therapy or are ineffective or not suitable for standard treatment;
4. Have at least one extracranial measurable lesion according to RECIST 1.1 criteria;
5. Estimated survival ≥ 12 weeks;
6. Baseline ECOG (Eastern Cooperative Oncology Group) score ≤ 1 point;
7. The patient has recovered from the toxicity of the prior treatment, i.e., CTCAE toxicity grade < 2 (unless the abnormality is related to the tumor or is stable as judged by the investigator and has little impact on safety or efficacy);
8. Venous access could be established; without contraindications of apheresis.

Exclusion Criteria:

1. Patients with prior or current other malignancies;
2. Presence of brain metastases and clinically significant central nervous system disease;
3. Prior antitumor therapy (prior to blood collection for CAR-T preparation) : targeted therapy, epigenetic therapy, or investigational drug therapy within 14 days or at least 5 half-lives, whichever is shorter;
4. Subjects with positive HBsAg or HBcAb positive and peripheral blood HBV DNA titer is higher than the lower limit of detection of the research institution; HCV antibody positive; HIV antibody positive; CMV DNA titer is higher than the lower limit of detection of the research institution; EBV DNA titer is higher than the lower limit of detection of the research institution
5. Those who have a positive sputum smear and T-cell test for tuberculosis infection;
6. Patients with objective evidence of a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, and severe impairment of lung function, both past and present;
7. Patients have a severe allergic history;
8. Patients with severe heart disease or uncontrollable refractory hypertension;
9. Patients with severe liver and kidney dysfunction or consciousness disorders;
10. Active autoimmune or inflammatory diseases of the nervous system;
11. Uncontrolled infections that need antibiotics treatment;
12. Live attenuated vaccine within 4 weeks before screening;
13. Alcoholics or persons with a history of drug abuse;
14. Pregnant or Lactating Women; Patients and his or her spouse have a fertility plan within two years after CAR-T cell infusion;
15. Any unsuitable to participate in this trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | within 52 weeks post-infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome are graded by American Society for Transplantation and Cellular Therapy (ASTCT) criteria.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | within 52 weeks post-infusion
  The Objective Response Rate (ORR) is the percentage of participants who achieved Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Concentration of CAR-T cells | Days 2, 5, 8, 11, 14, 21, 28, 35 and weeks 6, 12, 18, 26, 34, 42, 52 after infusion
  Concentration of CAR-T cells measured by Flow cytometry after CAR-T infusion
Progression-free survival(PFS) | within 52 weeks post-infusion
  Progression-free survival(PFS) refers to the time from cell reinfusion to the first assessment of tumor progression or death from any cause.
Overall survival(OS) | within 52 weeks post-infusion
  Overall survival (OS) refers to the time from the time the patient received an infusion of CAR-T cells until death (from any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, MD, Principal Investigator — Principal Investigator Sanbin Wang 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- Sanbin Wang, Kunming, Yunnan, China